CLINICAL TRIAL: NCT01463371
Title: Effects of Long-Term Azithromycin Treatment on Airway Oxidative Stress Markers in Patients With Stable Non-Cystic Fibrosis Bronchiectasis
Brief Title: Effects of Azithromycin on Airway Oxidative Stress Markers in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Sociedad Valenciana de Neumología (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 04/2004/0144
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2011-10

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Oxidative stress markers; Airway inflammation
MeSH Terms: conditions — Bronchiectasis | interventions — Azithromycin; Aftercare

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): without azithromycin
- azithromycin (Active Comparator): treatment with azithromycin during three months
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 250 mg three times a week during three months
  Other Names: Before treatment or after treatment
  Arms: azithromycin

SUMMARY:
The mechanism by which macrolide antibiotics have immune modifying effects independent from its antibacterial activity has not been well established. In the present work, the investigators will analyze the effect of long-term treatment with azithromycin (250 mg three times per week during three months) on airway oxidative stress markers in exhaled breath condensate of adult patients with stable non-CF bronchiectasis.

DETAILED DESCRIPTION:
The mechanism by which macrolide antibiotics have immune modifying effects independent from its antibacterial activity has not been well established. In the present work, we will analyze the effect of long-term treatment with azithromycin (AZ) on airway oxidative stress markers in exhaled breath condensate of adult patients with stable non-CF bronchiectasis. Patients will be randomized in an open label model to receive AZ 250 mg three times per week during three months or nothing.Dyspnea (Borg scale), exacerbations (Nº) in the last three months, sputum volume (cc), sputum colour (15-point scale), and health related quality of life (Questionnaire St.George) will be measured in both groups before and after treatment. Lung function, sputum culture, CT scan (Bhalla score) and inflammatory markers in blood (ESR, PCR),exhaled air (Nitric Oxide,) and exhaled condensed air (pH, nitrites, isoprostane) will be assessed before and after treatment. Relationships between clinical and inflammatory markers will be studied

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of bronchiectasis based on lung HRCT and clinical symptoms
* Clinically stable in previous four weeks without exacerbations
* Informed consent

Exclusion Criteria:

* Bronchiectasis secondary to Cystic fibrosis, pulmonary surgical processes, immune deficiency, emphysema, allergic bronchopulmonary aspergillosis or diffuse interstitial pulmonary diseases
* Intolerance to macrolides or severe liver disease.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Changes in Nitric oxide,8-isoprostane, pH, nitrites (NO2) and nitrates(NO3) in exhaled breath condensate. | Before and after three months of treatment
  Oxidative stress and NO metabolism in airway were investigated by measuring pH and the concentration of 8-isoprostane, nitrites (NO2-) and nitrates (NO3-) in EBC. Exhaled NO was also determined in all patients.

SECONDARY OUTCOMES:
Number of Exacerbations | Before and after three months of treatment
  exacerbations was defined by hospital admissions or antibiotics prescription
changes in lung function | Before and after three months of treatment
  Changes in FEV1, FVC.
colour and volume sputum, | Before and after three months of treatment
  In order to analyze sputum characteristics, three sterile containers were given to collect all sputum produced during three consecutive days. The average of the three days was calculated and expressed in mL/day. Sputum colour was scored using a scale developed and validated in our laboratory, which ranged from zero to fifteen: transparent (0), white (1), progressive intensities of yellow (2-7), green (8-10) and brown (10-15). Colour scores were decided after agreement between two investigators
Impact on functional capacity and health related quality of life | Before and after three months of treatment
  The impact on functional capacity and patient´s daily life was evaluated with the Medical Research Council Dyspnea scale (MRC) and the Spanish version of the Saint George's respiratory questionnaire of quality of life (SGRQ)
Changes in HRCT Lung scores | Before and after three months of treatment
  Standard lung HRCT scan was performed to quantify the extension of bronchiectasis

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo De Diego Damia, MD, Principal Investigator — Instituto Investigación Sanitaria La Fe
Locations (1):
- University Hospital La Fe, Valencia, Spain